CLINICAL TRIAL: NCT01037907
Title: A Placebo-controlled Phase IIa Study of Orally Administered BGC20-0134/Pleneva TM (Structured Lipid) in Patients With RRMS
Brief Title: A Study of Orally Administered BGC20-0134 (Structured Lipid) in Patients With Relapsing Remitting Multiple Sclerosis (RRMS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BGC20-0134-02
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Oral treatment for MS; Oral drug for multiple sclerosis; Oral RRMS; Oral relapsing remitting multiple sclerosis; Gamma Linolenic Acid; GLA; Fatty acid; Triglyceride; Structured lipid; MRI; Magnetic resonance imaging; gadolinium enhancing lesions; expanded disability status scale; EDSS; Demyelination; Remyelination; TGFB1; Transforming growth factor beta 1; cytokines; disease modifying therapy; immunomodulator; Anti inflammatory; Pro inflammatory; TNF alpha; interleukin 1 beta; interferon gamma; Fayaz Master; Omega 6; Polyunsaturated fatty acid; Cytokine balance; Pleneva TM; BGC20-0134; RRMS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Demyelinating Diseases; Camurati-Engelmann Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BGC20-0134 (Pleneva TM) (Experimental): Structured lipid
  Interventions: Drug: Pleneva TM BGC20-0134
- Placebo control (Placebo Comparator): Placebo - dummy pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pleneva TM BGC20-0134 — Placebo or 5 g dose
  Arms: BGC20-0134 (Pleneva TM)
Drug: Placebo — Placebo or 5 g dose
  Arms: Placebo control

SUMMARY:
To determine the efficacy and safety of an oral drug (BGC20-0134) in patients with relapsing remitting multiple sclerosis. Specifically, the cumulative number of new gadolinium enhancing lesions after 24 weeks of treatment with BGC20-0134.

DETAILED DESCRIPTION:
Primary outcome measure:

The cumulative number of new GdE T1 lesions developing while on treatment.

Secondary outcome measures:

* MRI:

  * Cumulative number of total GdE T1 lesions developing while on treatment
  * Cumulative number of new T2 lesions
  * Patients free of GdE (T1-weighted) lesions at week 24
  * Change in volume of GdE T1
  * Brain atrophy
  * Cumulative number of new T1 hypointense lesions (black holes)
* Disease burden, T1 and T2 lesion activity at week 48.
* Number of clinical relapses from baseline to the end of treatment. • Change on the Expanded Disability Status Scale (EDSS)
* Number of patients requiring methylprednisolone treatment for a relapse.
* Serum levels of pro- and anti-inflammatory cytokines.
* Quality of life (MSQOL-54)

Eligibility Criteria

MS-Related inclusion criteria

1. Diagnosis of relapsing MS according to the revised 2005 McDonald criteria.
2. Has shown disease activity defined by 1 or more MS attack within the last year which has been documented in prior medical notes and or the presence of active lesions on historical scans being either (based on radiology report or investigator review of MRI):

   1. Gd-enhancing on any scan obtained in the last year, or
   2. new T2 lesions between two scans both obtained within the last year.
   3. A minimum total of 9 T2 lesions reported on a recent MRI obtained within 1 month prior to the screening visit.
3. Baseline EDSS score 0 - 5.5.
4. Has refused to be treated with approved disease modifying therapies available for MS, for any reason and once the investigator has fully informed the patient about the related benefits and potential adverse events associated with such treatments. Also, patients for whom such treatments have proved to be intolerable.

Exclusion Criteria:

1. Has experienced an MS relapse or received systemic corticosteroids or adrenocorticotropic hormone (ACTH) in the previous 1 month.
2. Has a secondary progressive (SPMS), progressive relapsing (PRMS), or primary progressive MS (PPMS).
3. Has received any of the following agents to treat MS (approved or unapproved):

   * Within the previous 3 months: interferon beta, glatiramer acetate, intravenous immunoglobulin or plasmapheresis.
   * Within the previous 12 months: natalizumab, daclizumab, cytapheresis, azathioprine, cladribine, cyclophosphamide, methotrexate, mitoxantrone, mycophenolate, pixantrone, sirolimus, tacrolimus, or other agents typically used to prevent transplant rejection or as cancer chemotherapy, excluding hormonal treatments.
   * Ever having received: stem cell or bone marrow transplant, total lymphoid irradiation, vaccine therapy for MS, or monoclonal antibodies whose effects may be longer than 1 year (such as alemtuzumab or rituximab).
   * Within the previous 3 months: any other agents given for the non-symptomatic treatment of MS which are not included above, including over-the-counter, herbal and nutritional supplements. However, if the agent is being taken primarily to treat another medical condition, then it is allowed as long as the dose is unchanged within the previous 3 months and is unlikely to change before week

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing MS according to the revised 2005 McDonald criteria
* Has shown disease activity defined by 1 or more MS attack within the last year which has been documented in prior medical notes and or the presence of active lesions on historical scans being either (based on radiology report or investigator review of MRI):
* Gd-enhancing on any scan obtained in the last year, or
* new T2 lesions between two scans both obtained within the last year
* A minimum total of 9 T2 lesions reported on a recent MRI obtained within 1 month prior to the screening visit
* Baseline EDSS score 0 - 5.5
* Has refused to be treated with approved disease modifying therapies available for MS, for any reason and once the investigator has fully informed the patient about the related benefits and potential adverse events associated with such treatments. Also, patients for whom such treatments have proved to be intolerable

Exclusion Criteria:

* Has experienced an MS relapse or received systemic corticosteroids or adrenocorticotropic hormone (ACTH) in the previous 1 month
* Has a secondary progressive (SPMS), progressive relapsing (PRMS), or primary progressive MS (PPMS).
* Has received any of the following agents to treat MS (approved or unapproved):
* Within the previous 3 months: interferon beta, glatiramer acetate, intravenous immunoglobulin or plasmapheresis
* Within the previous 12 months: natalizumab, daclizumab, cytapheresis, azathioprine, cladribine, cyclophosphamide, methotrexate, mitoxantrone, mycophenolate, pixantrone, sirolimus, tacrolimus, or other agents typically used to prevent transplant rejection or as cancer chemotherapy, excluding hormonal treatments
* Ever having received: stem cell or bone marrow transplant, total lymphoid irradiation, vaccine therapy for MS, or monoclonal antibodies whose effects may be longer than 1 year (such as alemtuzumab or rituximab)
* Within the previous 3 months: any other agents given for the non-symptomatic treatment of MS which are not included above, including over-the-counter, herbal and nutritional supplements. However, if the agent is being taken primarily to treat another medical condition, then it is allowed as long as the dose is unchanged within the previous 3 months and is unlikely to change before week 24.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2009-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The cumulative number of new gadolinium-enhanced (GdE) T1 weighted lesions developing while on treatment (specifically the sum of new GdE T1 lesions seen on MRI at weeks 12, 16, 20 and 24). | 24 weeks

SECONDARY OUTCOMES:
Cumulative number of total GdE T1 weighted lesions developing while on treatment | 24 weeks
Cumulative number of new T2 weighted lesions | 24 weeks
Patients free of GdE (T1-weighted) lesions | 24 weeks
Change in volume of GdE T1 weighted lesions | 24 weeks
Change in volume of T2 lesions | 24 weeks
Brain atrophy | 24 weeks
Cumulative number of new T1 hypointense lesions (black holes) | 24 weeks
Disease burden, T1 and T2 lesion activity at week 48. | 48 weeks
Number of clinical relapses from baseline during the first 24 weeks. | 24 weeks
Change on the Expanded Disability Status Scale (EDSS) during the first 24 weeks | 48 weeks
Number of patients receiving methylprednisolone treatment for a relapse during the first 24 weeks. | 48 weeks
Serum levels of cytokines during the first 24 weeks. | 24 weeks
Quality of life (MSQOL-54) assessment | 48 weeks
PK for determination of circulating levels of BGC20-0134 and plasma concentrations of dihomo-gamma linolenic acid (DHGLA) during the first 24 weeks. | 24 weeks
Overall safety of BGC20-0134 | 48 weeks

CONTACTS AND LOCATIONS:
Locations (35):
- Belgium (3):
  - University Hospital Gent, Ghent
  - AZ St. Jan Brugge Oostende AV., Ruddershove
  - AZ ALMA, Sijsele
- France (4):
  - CHU Amiens-Hôpital Nord-, Amiens
  - CHU Clermont Ferrand-Hôpital Gabriel Montpied-, Clermont
  - CHRU Strasbourg- Hôpital Civil-1 place de l'hôpital, Strasbourg
  - CHU Toulouse-Hôpital Purpan, Toulouse
- Germany (11):
  - Klnik Hohe Warte, Bayreuth
  - Jüdisches Krankenhaus Berlin, Berlin
  - Universitätsklinikum Charité, Campus Mitte, Berlin
  - Klinikum der Ruhr-Universität Bochum, Bochum
  - Universitätsklinikum der Heinrich-Heine-Universität Düsseldorf, Düsseldorf
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Magdeburg A.ö.R, Magdeburg
  - Klinikum Osnabrück Klinik für Neurologie, Osnabrück
  - Universitätsklinikum Rostock AöR, Rostock
  - Neurologische und psychiatrische Praxis, Stuttgart
  - Universitätsklinikum Ulm, Ulm
- Poland (4):
  - Medical University of Gdansk Ul. Nowe Ogrody 1-6, Gdansk
  - Upper Silezian Medical Center SAM Ul Ziolowa 45/47, Katowice
  - Medical University of Lodz, Lodz
  - Samodzielny Publiczny Szpital Kliniczny, Lublin
- Russia (6):
  - State Medical University named after I.P. Pavlov, Saint Petersburg, Str. L. Tolstogo 6/8
  - City hospital # 11 Str. Dvintcev 6, Moscow
  - Moscow regional institute of clinical research named after M.F. Vladimirsky, Moscow
  - Institute of Human Brain, str. Acad. Pavlov, St-Petersburg, Saint Petersburg
  - City hospital # 9 Str. B. Gornaya 43, Saratov, Saratov
  - hospital # 33 pr. Lenina 54, Nizniy Novgorod, Veliky Novgorod
- Spain (7):
  - Hospital Universitari de Girona, Girona, Avda.De Franca, S/n
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Vall'd Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Ntra Sra de la Candelaria, Santa Cruz de Tenerife

REFERENCES:
- See also: Sponsor's website — http://www.btgplc.com